CLINICAL TRIAL: NCT05781906
Title: Single-center, Open-label, Multi-dose Study to Investigate the Human Mass Balance in Healthy Adult Male Following Multiple Oral Doses of HMPL-523 Tablets Followed by a Single Oral Dose of 300 mg/150 µCi [14C]HMPL-523 Suspension
Brief Title: Human Mass Balance of [14C]HMPL-523 in Healthy Adult Male Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-523-00CH3
Record Dates: First submitted 2023-02-07; First posted 2023-03-23 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Imumune Thrombocytopenia(ITP) Human Mass Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HMPL-523 (Experimental): HMPL-523 Tablet 300 mg QD7 days followed by a single oral dose of [14C]HMPL-523 suspension
  Interventions: Drug: HMPL-523; Drug: 150 µCi [14C]HMPL-523

INTERVENTIONS:
Drug: HMPL-523 — D1-D7: HMPL-523 Tablet 300 mg QD
  Other Names: HMPL-523 tablets
Drug: 150 µCi [14C]HMPL-523 — D8: [14C] HMPL-523 Suspension 300 mg/150 μCi Single dose
  Other Names: 150 µCi [14C]HMPL-523 suspension under fed condition

SUMMARY:
To evaluate the absorption, metabolism and excretion of HMPL-523 in healthy male Chinese subjects following multiple oral doses of HMPL-523 tablets followed by a single oral dose of [14C]HMPL-523 suspension

DETAILED DESCRIPTION:
a single-center, non-randomized, open-label, human mass balance, phase 1 study to evaluate the absorption, metabolism and excretion following multiple oral doses of HMPL-523 tablets, followed by a single oral dose of 300 mg/150 µCi [14C]HMPL-523 suspension in healthy adult male Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have voluntarily participated in the study and signed the informed consent form with good compliance;
2. Healthy male subjects aged 18-40 years (inclusive);
3. Subjects weighing ≥ 50 kg
4. Subjects in good health status

Exclusion Criteria:

1. Subjects with a history of gastrointestinal surgery, renal surgery, cholecystectomy and other procedures that in the judgment of the investigator may affect drug absorption or excretion
2. hypersensitivity to the investigational product and its excipients
3. Subjects with diseases affecting the absorption, distribution, metabolism and excretion of oral drugs,
4. Subjects with fear of needles, hemophobia, difficulty collecting venous blood, or special requirements for diet, who cannot comply with uniform diet
5. Subjects who are abnormal with clinical significance for C-reactive protein or positive for coronavirus nucleic acid detection in coronavirus infection screening
6. Subjects who have participated in another clinical trial of other drugs and have received such investigational product within 3 months prior to the first dose
7. Having any other diseases or conditions that may affect the normal performance of the study or the evaluation of the study data, or having other conditions that are not suitable for the study, as judged by investigators

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
the Human Mass Balance | Day1-Day7
  To evaluate the absorption, metabolism and excretion of HMPL-523 in healthy male Chinese subjects following multiple oral doses of HMPL-523 tablets
the Human Mass Balance | Day8
  To evaluate the absorption, metabolism and excretion of HMPL-523 in healthy male Chinese subjects followed by a single oral dose of [14C]HMPL-523 suspension

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, Principal Investigator — offices director
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR